CLINICAL TRIAL: NCT00643396
Title: Phase II Trial of Consolidative Thoracic Radiotherapy for Extensive Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: LU-23929/23929
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2012-04

CONDITIONS: Extensive Stage Small Cel Lung Cancer
Keywords: small cell lung cancer; radiotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma

INTERVENTIONS:
Radiation: thoracic radiotherapy

SUMMARY:
The majority of patients with small cell lung cancer have incurable extensive stage disease. The usual initial treatment for this condition is chemotherapy which produces responses in about 50-80% of patients. Despite this, the cancer usually returns. Once common body region where it re-grows is in the chest, which can cause symptoms such as shortness of breath, cough, difficulty swallowing, pain and bleeding. These symptoms can worsen a patient's quality of life and in some situation be life-threatening. In this study , we propose to give patients who have extensive stage small cell lung cancer which responds to chemotherapy radiotherapy treatments to the chest. By giving this type of radiation before the cancer has a chance to re-grow, we hope to control the disease within the chest and prevent future symptoms that it may cause if the cancer were to re-grow in the chest. Patients treated on the protocol will be checked regularly for disease control, quality of life and radiation side effects, if any.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmation of small cell lung cancer
* extensive stage disease
* adequate pulmonary function tests (FEV-1>1.0, DLCO>50%)
* patients of childbearing potential must practice adequate contraception
* age ≧ 18 years
* Karnofsky performance status ≧ 70
* documented objective response to initial chemotherapy
* signed study-specific informed consent form

Exclusion Criteria:

* complete or subtotal tumor resection
* non-small cell histology
* prior or concurrent malignancy except non-melanoma skin cancer unless disease-free for at least 5 years
* prior chest or neck RT
* inadequate pulmonary function tests (FEV-1<1.0 OR DLCO<50%)
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
local control | we anticipate completing accrual to the study in 12 months with most local failure events occuring within 2 years of treatment

SECONDARY OUTCOMES:
radiotherapy toxicities | 1-2 years after study treatment
patient quality of life | 1-2 years after study treatment
overall survival | 1-2 years after study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Don Yee, MD, FRCPC, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada